CLINICAL TRIAL: NCT04631887
Title: The Feasibility Study of The Delivery of The Book From Self Help Plus: "Doing What Matters in Times of Stress: An Illustrated Guide"
Brief Title: The Delivery of "Doing What Matters in Times of Stress: An Illustrated Guide"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Ceren Acarturk, Associate Professor, Koç University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020.200.IRB3.080
Record Dates: First submitted 2020-11-07; First posted 2020-11-17 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Stress; Quality of Life; Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: Doing What Matters in Times of Stress: An Illustrated Guide (Experimental): The intervention arm will receive the assigned intervention for five weeks. They will receive the intervention materials and will be called by psychologists three times (at the beginning, middle and end) during the intervention.
  Interventions: Behavioral: Doing What Matters in Times of Stress: An Illustrated Guide
- Control Arm: Wait List (No Intervention): The control arm has no intervention. The participants in the control arm will receive the intervention after the post-assessments are completed.

INTERVENTIONS:
Behavioral: Doing What Matters in Times of Stress: An Illustrated Guide — The "Doing What Matters in Times of Stress: An Illustrated Guide" is a booklet that is developed by World Health Organization. It is a stress management booklet formed to provide people skills for coping with stress and adversity. The booklet has accompanying audio exercises.
  Arms: Intervention Arm: Doing What Matters in Times of Stress: An Illustrated Guide

SUMMARY:
The feasibility study for the delivery of the "Doing What Matters in Times of Stress: An Illustrated Guide" will be carried out for Turkish and Syrian individuals with psychological stress. This feasibility study's sample will be adult Turkish and the Syrian refugees. The informed consent form and screening questionnaire of the feasibility study will be sent to the participants who have given this approval and 128 (64 Turkish and 64 Syrian) participants who meet the inclusion criteria will be included in the feasibility study. The psychological problems will be measured twice, before and after the intervention.

DETAILED DESCRIPTION:
Studies about the impact of epidemics such as Severe acute respiratory syndrome (SARS) on the psychological health of individuals show that psychological problems have been observed in individuals who are affected by the epidemic. Today, studies on the effects of COVID-19 on psychological health are also available in the literature, and the results of these studies are in line with those of previous studies on epidemics.

The aim of this project is to deliver the "Doing What Matters in Times of Stress: An Illustrated Guide" that is developed by the World Health Organization within Self Help Plus (SH+) intervention to decrease their psychological problems for a feasibility study. The feasibility study for the delivery of the SH+ book will be carried out and the psychological problems of the participants will be measured twice, before and after the intervention to evaluate the results.

The most important contribution of the Project is conducting a feasibility study with the "Doing What Matters in Times of Stress: An Illustrated Guide" which will be adapted to the Turkish culture based on the determination of Turkey's current psychological status, provide a form of intervention to the Turkish psychological intervention literature and to improve the psychological status of the participants in this project.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or above
* Being literate
* Being a Turkish citizen or a Syrian refugee
* Scoring 15 or above on Kessler Psychological Distress Scale (K10)

Exclusion Criteria:

* Imminent suicidal risk
* Being illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Change of the Patient Health Questionnaire-9 (PHQ-9) over time | Change from baseline (1 week before the intervention) to post assessment (6 weeks after the pre-assessment)
  Patient Health Questionnaire-9 is a 9 item questionnaire that aims to measure the severity of depression symptoms. Each of the 9 items are scored as "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score. Higher scores indicate decreased functional status and increased symptom-related difficulties.

SECONDARY OUTCOMES:
Change of the General Anxiety Disorder-7 (GAD-7) over time | Change from baseline (1 week before the intervention) to post assessment (6 weeks after the pre-assessment)
  General Anxiety Disorder-7 is a 7-item questionnaire that aims to measure anxiety symptoms. Each of the 7 items are scored as 0, 1, 2, and 3 to the response categories (0 = "not at all," to 3= "nearly every day"). The total score for the seven items ranges from 0 to 21. Higher scores indicate higher levels of anxiety.
Change of the PTSD Checklist for The Diagnostic and Statistical Manual of Mental Disorders 5 (DSM 5) (PCL-5) over time | Change from baseline (1 week before the intervention) to post assessment 6 weeks after the pre-assessment)
  The PTSD Checklist for DSM-5 is a 20-item questionnaire that assesses the symptoms of PTSD. In this study, a single question from each criteria of PTSD will be used. Overall four questions from PCL-5 will be assessed. Each of the 4 items are scored as 0, 1, 2, 3 and 4 (0 = "Not at all" to 4 = "Extremely"). The total score for the four items ranges from 0 to 16. Higher scores indicate higher levels of PTSD symptoms.
Change of the The World Health Organization Quality of Life (WHOQOL) over time | Change from baseline (1 week before the intervention) to post assessment 6 weeks after the pre-assessment)
  The World Health Organization Quality of Life questionnaire assesses various domains of life which are physical health, psychological health, social relationships, and environment. In this study, a single question from the questionnaire will be used which will be about the general quality of life. The question is scored from 1 to 5 on a response scale (1 = "Not at all" to 5 = "Completely"). A higher score indicate higher quality of life.
Change of the The General Self-Efficacy Scale over time | Change from baseline (1 week before the intervention) to post assessment 6 weeks after the pre-assessment)
  The General Self-Efficacy Scale is a 10-item questionnaire that assesses the general sense of perceived self-efficacy. Each of the 10 items are scored as 1, 2, 3 and 4 on a response scale (1 = "Not at all true" to 4 = "Exactly true"). The total score for the four items ranges from 10 to 40. Higher scores indicate higher perceived general self-efficacy, lower scores indicate lower perceived general self-efficacy.
Change of the The Acceptance and Action Questionnaire (AAQ-2) over time | Change from baseline (1 week before the intervention) to post assessment 6 weeks after the pre-assessment)
  The Acceptance and Action Questionnaire is a 7-item questionnaire that assesses the psychological flexibility. Each of the 7 items are scored as 1, 2, 3, 4, 5, 6 and 7 on a response scale (1 = "Never true" to 7 = "Always true"). The total score for the four items ranges from 7 to 49. Higher total scores mean less flexibility, while lower total scores mean more flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Kurt, PhD, Study Chair — Koç University; Zeynep Ilkkursun, MA, Study Chair — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dong L, Bouey J. Public Mental Health Crisis during COVID-19 Pandemic, China. Emerg Infect Dis. 2020 Jul;26(7):1616-1618. doi: 10.3201/eid2607.200407. Epub 2020 Jun 21. PMID 32202993
- [Background] Epping-Jordan JE, Harris R, Brown FL, Carswell K, Foley C, Garcia-Moreno C, Kogan C, van Ommeren M. Self-Help Plus (SH+): a new WHO stress management package. World Psychiatry. 2016 Oct;15(3):295-296. doi: 10.1002/wps.20355. No abstract available. PMID 27717271
- [Background] Fledderus M, Bohlmeijer ET, Pieterse ME, Schreurs KM. Acceptance and commitment therapy as guided self-help for psychological distress and positive mental health: a randomized controlled trial. Psychol Med. 2012 Mar;42(3):485-95. doi: 10.1017/S0033291711001206. Epub 2011 Jul 11. PMID 21740624

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT04631887/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT04631887/ICF_001.pdf